CLINICAL TRIAL: NCT02762760
Title: A Prospective Phase I Study to Evaluate the Safety of a Single Intra-articular Injection of Ampion™ as a Treatment for Arthritis of the Basal Thumb Joint
Brief Title: AP-011 Study to Evaluate the Safety of a Single Intra-articular Injection of Ampion™ for Arthritis of the Basal Thumb Joint
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ampio Pharmaceuticals. Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AP-011
Record Dates: First submitted 2016-05-02; First posted 2016-05-05 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-10

CONDITIONS: Osteoarthritis of the Hand
MeSH Terms: interventions — aspartyl-alanyl-diketopiperazine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AMPION™ (Experimental): AMPION™, up to 3 mL, single intra-articular injection. Ampion is the ultrafiltrate of 5% HSA.
  Interventions: Biological: AMPION™
- Saline (Experimental): Saline placebo, up to 3 mL, single intra-articular injection. Saline used as the comparator is 0.9% Sodium Chloride
  Interventions: Biological: Saline

INTERVENTIONS:
Biological: AMPION™ — AMPION™, up to 3 mL, single intra-articular injection. Ampion is the ultrafiltrate of 5% HSA.
  Arms: AMPION™
Biological: Saline — Saline placebo, up to 3 mL, single intra-articular injection. Saline used as the comparator is 0.9% Sodium Chloride
  Arms: Saline

SUMMARY:
This study will evaluate the safety of an intra-articular injection of AMPION™ in adults with pain due to osteoarthritis of the basal thumb joint.

DETAILED DESCRIPTION:
A prospective phase I study to evaluate the safety of a single intra-articular injection of Ampion™ as a treatment for arthritis of the basal thumb joint.

Primary Objective is:

To evaluate the safety of Ampion™ (up to 3 mL) in comparison to saline placebo (up to 3 mL) when injected into the basal thumb joint.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent to participate in the study.
2. Willing and able to comply with all study requirements and instructions of the site study staff.
3. Male or female, 40 years to 85 years old (inclusive).
4. Radiographic evidence of Basal joint arthritis (Eaton-Littler classification, stages 1 through 4).
5. Pain associated with basal joint arthritis, defined as a score ≥ 4 as evaluated by the Australian-Canadian OA Index (AUSCAN)-numeric rating score (NRS, 0-10).

Exclusion Criteria:

1. As a result of medical review and screening investigation, the Principal Investigator considers the subject unfit for the study.
2. Previous Ampion™ injection.
3. A history of allergic reactions to human albumin (reaction to non-human albumin such as egg albumin is not an exclusion criterion).
4. A history of allergic reactions to excipients in 5% human albumin (N-acetyltryptophan, sodium caprylate).
5. Women who are currently pregnant or who could become pregnant.
6. Inflammatory or crystal arthropathies, acute fractures, history of aseptic necrosis, as assessed locally by the Principal Investigator.
7. Any other disease or condition interfering with the free use and evaluation of the index thumb for the duration of the trial (e.g., congenital defects, stricture).
8. Major injury to the index thumb within the 12 months prior to screening.
9. Any pharmacological or non-pharmacological treatment targeting OA started or changed during the 4 weeks prior to treatment or likely to be changed during the duration of the study.
10. Use of the following medications are exclusionary:

    * IA injected pain medications in the study thumb during the study;
    * Analgesics containing opioids;
    * NSAIDs (including but not limited to ibuprofen, aspirin, naproxen, diclofenac) acetaminophen is available as a rescue medication during the study from the provided supply;
    * Topical prescription treatment on osteoarthritis index thumb during the study;
    * Significant anticoagulant therapy (e.g., Heparin or Lovenox) during the study (treatment such as Aspirin in the cardio-protective dose (81mg) and Plavix are allowed);
    * Systemic treatments that may interfere with safety or efficacy assessments during the study;
    * Immunosuppressants;
    * Use of corticosteroids > 10 mg prednisolone equivalent per day (if ≤ 10 mg prednisolone, the dose must be stable, defined as chronic use of the same dose for at least 1 month).
11. Any human albumin treatment in the 3 months before randomization.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-05; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Safety will be evaluated from Baseline to Week 4. monitoring incidence of AEs, thumb exam, vitals, and concomitant medication use | Baseline to 4 weeks
  The Clinical safety of treatment on base of the thumb will be assessed by recording AEs at all in-clinic visits and the 24-hour, post-injection telephone contact call, by the results of the physical examination of the thumb joint and vital signs (at all in-clinic visits), and by recording prior and concomitant medications including start/stop dates, indication, dose and frequency (at 24 hour post-injection telephone contact call and all in-clinic visits).

CONTACTS AND LOCATIONS:
Overall Officials: David Bar-Or, MD, Study Director — Ampio Pharmaceuticals. Inc.
Locations (1):
- Ampio Pharmaceuticals, Englewood, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided